CLINICAL TRIAL: NCT05747508
Title: A Randomized, Double-Blind, Placebo-Controlled Dose Escalation Clinical Study to Assess the Safety and Efficacy of Pulsed Inhaled Nitric Oxide (iNO) in Subjects With Pulmonary Hypertension Associated With Pulmonary Fibrosis on Long Term Oxygen Therapy (Part 1 and Part 2)
Brief Title: A Study to Assess Pulsed Inhaled Nitric Oxide in Subjects With Pulmonary Hypertension Associated With Pulmonary Fibrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bellerophon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PULSE-PHPF-001 Phase 2
Record Dates: First submitted 2021-07-27; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Fibrosis; Pulmonary Hypertension
Keywords: Pulmonary Fibrosis (PF); Pulmonary Hypertension; Inhaled Nitric Oxide; iNO; Long Term Oxygen Therapy; Oxygen
MeSH Terms: conditions — Pulmonary Fibrosis; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Inhaled Nitric Oxide (iNO) (Active Comparator): Pulsed inhaled iNO30, 45 and 75 mcg/kg Ideal Body Weight (IBW)/hour (hr)
  Interventions: Combination Product: INOpulse®
- Placebo (Placebo Comparator): Pulsed inhaled N2, 99.999% gas
  Interventions: Combination Product: Placebo
- Long Term Follow Up (Active Comparator): Pulsed inhaled iNO30, 45 or 75 mcg/kg IBW/hr
  Interventions: Combination Product: Long Term Follow Up

INTERVENTIONS:
Combination Product: INOpulse® — Patients will be treated by means of an INOpulse® device using an INOpulse® nasal cannula
  Arms: Inhaled Nitric Oxide (iNO)
Combination Product: Placebo — Patients will be treated by means of an INOpulse® device using an INOpulse® nasal cannula
  Arms: Placebo
Combination Product: Long Term Follow Up — Patients will be treated by means of an INOpulse® device using an INOpulse® nasal cannula
  Arms: Long Term Follow Up

SUMMARY:
A randomized, double-blind, placebo-controlled dose escalation study to assess the safety and efficacy of pulsed, inhaled nitric oxide (iNO) in subjects with pulmonary fibrosis on long term oxygen therapy.

DETAILED DESCRIPTION:
A Phase 2b, randomized, double-blind, placebo-controlled dose escalation clinical study to assess the safety and efficacy of pulsed, inhaled nitric oxide in subjects with and without pulmonary hypertension associated with pulmonary fibrosis on long term oxygen therapy (Part 1 and Part 2)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with pulmonary fibrosis by high resolution CT scan performed in the 6 months prior to screening associated with one of the following conditions and confirmed using one of the following guidelines, as per American Thoracic Society (AGS) / European Respiratory Society (ERS) / Japanese Respiratory Society (JRS) / Latin American Thoracic Association (ALAT):

  * Major idiopathic interstitial pneumonias (IIPs) diagnosis or suspected as one of the following:

    * Idiopathic pulmonary fibrosis
    * Idiopathic nonspecific interstitial pneumonia
    * Respiratory bronchiolitis-interstitial lung disease
    * Desquamative interstitial pneumonia
    * Cryptogenic organizing pneumonia
    * Acute interstitial pneumonia
  * Rare IIPs diagnosis by one of the following:

    * Idiopathic lymphoid interstitial pneumonia
    * Idiopathic pleuroparenchymal fibroelastosis
  * Unclassifiable idiopathic interstitial pneumonias
  * Chronic hypersensitivity pneumonitis
  * Occupational lung disease
* Have been using oxygen therapy by nasal cannula for at least 4 weeks
* 6-Minute Walk Distance (6MWD) ≥ 100 meters and ≤ 450 meters at screening and Baseline/Randomization visits
* World Health Organization (WHO) Functional Class II-IV
* Forced Vital Capacity ≥ 40% predicated within the last 6 months prior to the screening run-in period
* Age between 18 and 85 years (inclusive)

Exclusion Criteria:

* Pregnant or breastfeeding females at Screening
* In the last 6 months prior to screening, evidence of any connective tissue disease with FVC > 60% unless there is evidence of moderate to severe fibrosis on CT scan in the opinion of the local radiologist/Investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of escalating doses of iNO in patient's life participation as assessed in minutes per day of moderate to vigorous activity. | Change from baseline to week 8 or 16
  Part 1 - Blinded Treatment Period

OTHER OUTCOMES:
Change in 6-minute walking test (6MWT) from baseline | Change from baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Difference in activity as measured using ActiGraph devices | Change from baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Percentage of patients with ≥15% decrease in activity | Change from baseline to to week 8 or 16
  Part 1 - Blinded Treatment Period
Difference in dyspnea as measured by University of California San Diego Shortness of Breath Questionnaire | Change from baseline to to week 8 or 16
  The University of California San Diego Shortness of Breath Questionnaire is a 24-item questionnaire developed to measure breathlessness associated with activities of daily living, on a scale between zero and five where 0 is not at all breathless and 5 is maximally breathless or too breathless to do the activity. The responses to all items are summed up to provide the overall score that can range from 0 (best outcome) to 120 (worst outcome).
Difference in St. George Respiratory Questionnaire and sub-groups | Change from baseline to to week 8 or 16
  St. George Respiratory Questionnaire and sub-groups is a tool for assessing quality of life that has previously been validated for the use with patients with interstitial lung disease. It is a responsive tool that has three domains: symptoms, activity and impact (on daily life)
Percentage of patients with a clinically meaningful difference (reduction of at least 4 points) in the disease-specific quality of life measured using the disease specific St. George Respiratory Questionnaire (SGRQ) | Change from baseline to to week 8 or 16
  Part 1 - Blinded Treatment Period
Change in N-terminal (NT)-ProBNP (absolute and percentage) | Change from baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Time to clinical improvement | Baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Time to clinical worsening | Baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Incidence and severity of treatment emergent adverse events, including those related to INOpulse® device deficiency | Baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Adverse events that may be due to rebound associated with a temporal acute withdrawal of investigational study drug | Baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Change in diffusing capacity of the lungs for carbon monoxide (DLCO) | Baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Mortality | Baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Hospitalization (all cause and for cardiopulmonary or other cause) | Baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Change in Forced Expiratory Volume at 1 minute (FEV1) | Baseline to week 8 or 16
  Part 1 - Blinded Treatment Period
Change in Forced Vital Capacity (FVC) | Baseline to week 8 or 16
  Part 1 - Blinded Treatment Period

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics
Locations (23):
- United States (23):
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - University of California, Los Angeles, California
  - University of California Davis Health, Sacramento, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Healthcare Pulmonary & Critical Care Research, Austell, Georgia
  - Loyola University, Chicago, Illinois
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - The Lung Research Center (St. Luke's), Chesterfield, Missouri
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Thomas Jefferson University Korman Respiratory Institute, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah Health Sciences, Salt Lake City, Utah
  - Inova Heart and Vascular Institute Advanced Lung Disease Clinic, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No